CLINICAL TRIAL: NCT04868825
Title: Safety and Efficacy Evaluation of the Ivory Dentin Graft Device - Long Term Follow-Up
Brief Title: Safety and Efficacy Evaluation of the Ivory Dentin Graft Device (IvoryGraft) - Long Term Follow-Up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ivory Graft Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QF-04-09-01P-
Record Dates: First submitted 2021-04-20; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Deficiency of Alveolar Ridge (Disorder); Alveolar Bone Grafting; Mandibular Prosthesis User
Keywords: Bone substitutes; Dental implants; Dentin

STUDY DESIGN:
Intervention Model Description: prospective, randomized, semi double blinded with blinded assessments study comparing patients grafted with Ivory Dentin Graft (study arm) and patients grafted with OsteoBiol Gen Os (control arm) for alveolar ridge preservation following tooth extraction.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the graft performing sub-investigator and the study coordinator are un-blinded to subjects allocation - semi double blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Intervention) (Experimental)
  Interventions: Device: Ivory Dentin Graft
- Active Comparator (Active Comparator)
  Interventions: Device: OsteoBiol Gen-Os

INTERVENTIONS:
Device: Ivory Dentin Graft — Ivory Dentin Graft is a bone graft material for the repair or augmentation of bone defects in dental procedures. It consists of sterile 300 - 900 μm porous particles or granules of hydroxyapatite and collagen which retain the natural form of the source porcine dentin and protein matrix. (Packed Vial: 1.00 gr; Packed Syringe: 1.0 gr)
  Arms: Experimental (Intervention)
Device: OsteoBiol Gen-Os — Comparator control device A natural porcine origin cortico-cancellous heterologous bone mix consists of sterile 250 - 1000 μm porous particles of hydroxyapatite and collagen (Packed Vial: 1.0 gr)
  Arms: Active Comparator

SUMMARY:
long-term safety and performance of Ivory Dentin Graft. Ivory Dentin Graft is at least as good as the competitor treatment group (OsteoBiol Gen-Os) for alveolar ridge preservation following tooth extraction.

DETAILED DESCRIPTION:
This clinical investigation is part of the post-market development process of the investigational device of Ivory Graft Ltd. in order to satisfactory validate the safety, tolerability and effectiveness of Ivory Dentin Graft as required by the sponsor's European Union (EU) notified body.

The clinical Investigation was conducted with the stated confirmation applying European regulations; International Conference of Harmonization - Good Clinical Practice (ICH-GCP) guidelines, ISO 14155:2011, and with a relevant subject population for the study objectives. Israeli Ministry of Health registration Number: 20173907.

The purpose of this investigation is to evaluate the safety, tolerability and effectiveness of Ivory Dentin Graft for long-term evaluations, compared to the active comparator, OsteoBiol-Gen-Os® graft, as a treatment for alveolar ridge preservation following tooth extraction.

Long term follow-up: from completion of visit 5 (implant placement) up to 5 years from bone grafting per subject (visits 6-9).

Study design: A prospective, randomized, semi double-blinded with blinded assessments clinical investigation, comparing between subjects grafted with Ivory Dentin Graft (Investigational group) and subjects grafted with OsteoBiol-Gen-Os® (comparator group)

Study population: A total of 41 male and female adult subjects between the ages of 18 to 80 years old requiring alveolar ridge preservation that already had mandibular premolar or molar tooth extraction were included to this ongoing study (NCT03150472; short-term follow-up of 4 months following grafting was completed on September 9, 2020). Twenty-three (23) were previously randomized and grafted with Ivory Dentin Graft (Investigational group) and 18 with the active comparator, OsteoBiol Gen-Os (Comparator group). Five (5) subjects early withdrawn the short-term study resulting in 36 subjects included for this long-term study.

Sample size Justification and Statistical Analysis Plan: The rationale for sample size calculation is based on demonstrating non-inferiority in the study primary endpoint between the investigational and the reference comparator groups. The calculations assume a difference of up to 30% (percent as in unit of measure and not of relative difference) woven bone between the treatments, which will be considered equivalent (non-inferiority) and standard deviation of 32%.

Intended Use: bone graft material for the repair or augmentation of bone defects in dental procedures.

Clinical Follow-up: subjects are medically monitored for any long-term side effects (6 and 10 months, 2.5 and 5 years following their grafting procedure) and their dental condition is also followed by dental hygienist.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient 18 up to 80 years.
2. Patient requiring at least one implant placement following mandibular pre-molar or molar tooth extraction.
3. Alveolar mandibular ridge (empty socket):

   * Height: not less than 10 mm, from the gingival margin to the mandibular nerve canal - as seen in the screening CT scan.
   * Width: not less than 5 mm, from buccal to lingual cortical plates - as seen in the screening CT scan.
4. Ability to give informed consent for the study by patient or legal guardian.
5. Willingness to undergo 7 follow up visits: 1 week, 1, 4, 6 and 10 months, 2.5 years and 5 years following dental graft implantation, as well as unscheduled sick visits.

   Exclusion Criteria:
6. Pregnancy (all women of childbearing age would be questioned and told by the consenting physician regarding that criteria).
7. Known or suspected hypersensitivity to the constituents of the bone graft material (for example porcine collagen)
8. Pathologies or conditions contraindicating surgery or presenting with active acute or chronic infections excluding periapical granuloma (for example osteomyelitis, sinusitis), uncontrolled diabetes
9. Immunologic disorders or autoimmune pathologies, in particular elderly
10. Serious bone diseases of endocrine aetiology
11. Serious disturbances of bone metabolism
12. Ongoing treatment with gluco- or mineralocorticoids, or with agents affecting calcium metabolism (e.g. calcitonin, bisphosphonates)
13. Irradiation therapy, chemotherapy or immunosuppressive therapy in the last 5 years
14. Malignancies
15. Severe Parafunction (bruxism and clenching)
16. Poor oral hygiene or active periodontitis
17. Heavy tobacco smoking habit (> 10 cigarettes per day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Success of implant placement in a rigid post grafting site | 5 years after grafting
  defined by dental implant survival
Number of Participants with Treatment-Related Adverse Events | 5 years after grafting
  through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Tal Lavi, PhD, Study Director — Ivory Graft Ltd.
Locations (1):
- Assaf HaRofeh Medical Center, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not intended to be shared as this will be a single site study. The study will be public at ClinicalTrial.gov

REFERENCES:
- [Background] Hansson S, Halldin A. Alveolar ridge resorption after tooth extraction: A consequence of a fundamental principle of bone physiology. J Dent Biomech. 2012;3:1758736012456543. doi: 10.1177/1758736012456543. Epub 2012 Aug 16. PMID 22924065
- [Background] Horowitz R, Holtzclaw D, Rosen PS. A review on alveolar ridge preservation following tooth extraction. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):149-60. doi: 10.1016/S1532-3382(12)70029-5. PMID 23040345
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Chrcanovic BR, Albrektsson T, Wennerberg A. Bone Quality and Quantity and Dental Implant Failure: A Systematic Review and Meta-analysis. Int J Prosthodont. 2017 May/June;30(3):219-237. doi: 10.11607/ijp.5142. Epub 2017 Mar 20. PMID 28319206
- [Background] Herrmann I, Lekholm U, Holm S, Kultje C. Evaluation of patient and implant characteristics as potential prognostic factors for oral implant failures. Int J Oral Maxillofac Implants. 2005 Mar-Apr;20(2):220-30. PMID 15839115
- [Background] Barone A, Todisco M, Ludovichetti M, Gualini F, Aggstaller H, Torres-Lagares D, Rohrer MD, Prasad HS, Kenealy JN. A prospective, randomized, controlled, multicenter evaluation of extraction socket preservation comparing two bovine xenografts: clinical and histologic outcomes. Int J Periodontics Restorative Dent. 2013 Nov-Dec;33(6):795-802. doi: 10.11607/prd.1690. PMID 24116363
- [Background] Mahesh L, Venkataraman N, Shukla S, Prasad H, Kotsakis GA. Alveolar ridge preservation with the socket-plug technique utilizing an alloplastic putty bone substitute or a particulate xenograft: a histological pilot study. J Oral Implantol. 2015 Apr;41(2):178-83. doi: 10.1563/AAID-JOI-D-13-00025. Epub 2013 Jun 17. PMID 23772806
- [Background] Lai VJ, Michalek JE, Liu Q, Mealey BL. Ridge preservation following tooth extraction using bovine xenograft compared with porcine xenograft: A randomized controlled clinical trial. J Periodontol. 2020 Mar;91(3):361-368. doi: 10.1002/JPER.19-0211. Epub 2019 Aug 23. PMID 31380563
- [Background] Pang C, Ding Y, Zhou H, Qin R, Hou R, Zhang G, Hu K. Alveolar ridge preservation with deproteinized bovine bone graft and collagen membrane and delayed implants. J Craniofac Surg. 2014 Sep;25(5):1698-702. doi: 10.1097/SCS.0000000000000887. PMID 25148644
- [Background] Jung RE, Sapata VM, Hammerle CHF, Wu H, Hu XL, Lin Y. Combined use of xenogeneic bone substitute material covered with a native bilayer collagen membrane for alveolar ridge preservation: A randomized controlled clinical trial. Clin Oral Implants Res. 2018 May;29(5):522-529. doi: 10.1111/clr.13149. Epub 2018 Apr 1. PMID 29607553
- [Background] Meloni SM, Tallarico M, Lolli FM, Deledda A, Pisano M, Jovanovic SA. Postextraction socket preservation using epithelial connective tissue graft vs porcine collagen matrix. 1-year results of a randomised controlled trial. Eur J Oral Implantol. 2015 Spring;8(1):39-48. PMID 25738178
- [Background] Lee JS, Cha JK, Kim CS. Alveolar ridge regeneration of damaged extraction sockets using deproteinized porcine versus bovine bone minerals: A randomized clinical trial. Clin Implant Dent Relat Res. 2018 Oct;20(5):729-737. doi: 10.1111/cid.12628. Epub 2018 Jul 27. PMID 30051954